CLINICAL TRIAL: NCT04656912
Title: Effect of Hyperbaric Oxygen Therapy Initiation Time in Acute Carbon Monoxide Poisoning
Brief Title: Hyperbaric Oxygen Therapy Initiation Time in Acute Carbon Monoxide Poisoning
Status: Completed | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Yong Sung Cha, Assistant Professor, Wonju Severance Christian Hospital
Other Study IDs: CO-HBO
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Hyperbaric Oxygenation; Carbon Monoxide Poisoning; Time
MeSH Terms: conditions — Carbon Monoxide Poisoning | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute CO poisoning: A diagnosis of CO poisoning was made according to medical history and carboxyhemoglobin >5% (>10% in smokers).
  Interventions: Procedure: Hyperbaric oxygen therapy

INTERVENTIONS:
Procedure: Hyperbaric oxygen therapy — Patients with any symptoms and signs were treated with HBO2. During the first HBO2, initial compression was performed to 2.8 atmospheres absolute (ATA) for 45 min, followed by 2.0 ATA for 60 min. If an additional HBO2 was possible within 24 h, then 2.0 ATA was administered for 90 min. Moreover, if necessary, patients were treated with HBO2, even after 24 h, until all symptoms resolved.

SUMMARY:
Hyperbaric oxygen therapy (HBO2) is recommended for symptomatic patients within 24 h of carbon monoxide (CO) poisoning. However, previous major studies found significantly better outcomes with HBO2 in patients treated within 6 h. Currently, there is no consensus on a CO poisoning-to-HBO2 interval that would not be beneficial.

Therefore, the investigators aimed to evaluate the difference in therapeutic effect depending on the poisoning-to-HBO2 interval after CO exposure in patients with acute CO poisoning who received HBO2 within 24 h. The investigators compared the neurocognitive outcomes of patients according to HBO2 time intervals based on the outcomes of patients treated within 6 h (control group) with propensity score matching using the CO poisoning registry of our hospital.

DETAILED DESCRIPTION:
In the United States, 50,000 patients with carbon monoxide (CO) poisoning are admitted to the hospital emergency departments annually, resulting in 1,500 deaths. CO poisoning can have serious neurologic sequelae. Immediate treatment, within 24 h after poisoning, is a reasonable recommendation for patients with CO poisoning. Most physicians do not treat with hyperbaric oxygen therapy (HBO2) 24 h after CO poisoning.

Weaver et al. conducted a double-blind randomized control trial (RCT) satisfying all Consolidated Standards for the Reporting of Trials guidelines, which showed that HBO2 significantly reduced the rate of cognitive sequelae than normobaric oxygen therapy (NBO2) 6 weeks and 12 months post-treatment in patients with acute symptomatic CO poisoning. Although the aforementioned study used a maximum poisoning-to-HBO2 interval of 24 h in the inclusion criteria, more than 60% of enrolled patients were treated with HBO2 in less than 6 h after CO poisoning and the mean poisoning-to-HBO2 time was 5.8 h. In addition, in a subgroup with poisoning-to-HBO2 interval > 6 h, the mean interval was 8.6 h. Therefore, their study results were actually powered to determine the benefit of HBO2 within 6 h post-CO poisoning; hence, it is unknown whether HBO2 reduces the neurocognitive sequelae occurrence rate if performed beyond 6-12 h from CO poisoning.

Currently, there is no consensus on a CO poisoning-to-HBO2 interval that would not be beneficial. Therefore, the investigators aimed to evaluate the difference in therapeutic effect depending on the poisoning-to-HBO2 interval after CO exposure in patients with acute CO poisoning who received HBO2 within 24 h. The investigators compared the neurocognitive outcomes of patients according to HBO2 time intervals based on the outcomes of patients treated within 6 h (control group) with propensity score matching to make tight adjustments to significant differences in patient baseline characteristics using the CO poisoning registry of our hospital.

The investigators classified the patients included in the study into two groups: an early group (≤ 6 h, control group) and a late group (6-24 h, case group), based on the time from patient rescue from CO source to the start of the first HBO2 session. In addition, patients who received HBO2 at 6-24 h were divided into case 1 group (> 6 h and ≤ 12 h) and case 2 group (≥ 12 h and ≤ 24 h), and outcomes were compared with those of patients who received HBO2 within 6 h from CO exposure. Moreover, the investigators classified poisoning severity based on the necessity for intubation; mildly and severely poisoned patients were defined as those not requiring and requiring intubation, respectively

ELIGIBILITY:
Inclusion Criteria:

* CO poisoned patients

Exclusion Criteria:

1. Not treated with HBO2
2. < 16 years old
3. Non-acute CO poisoning
4. Received HBO2 more than 24 h after poisoning
5. A history of previous stroke or neurocognitive diseases
6. Did not undergo follow-up until 6 months
7. Received specific treatment other than HBO2, such as therapeutic hypothermia
8. A history of previous CO exposure
9. A serious illness that can affect the patient's prognosis such as advanced cancer
10. A cardiac arrest before ED arrival
11. No recorded data on important variables, such as time from CO exposure to the start of first HBO2

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CO poisoned patients
Sampling Method: Probability Sample
Enrollment: 706 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Frequency of poor global deterioration scale (GDS) at 1 month after CO exposure in the overall matched cohort | At 1 month after CO exposure
  Frequency of poor GDS (4-7 scores) outcome at 1 month after CO exposure between early group and late group
  *GDS (the minimum and maximum: 1-7, higher scores mean a worse outcome) Poor GDS outcome means from 4 to 7 in GDS score.
Frequency of poor GDS at 6 months after CO exposure in the overall matched cohort | At 6 months after CO exposure
  Frequency of poor GDS outcome at 6 months after CO exposure between early group and late group

SECONDARY OUTCOMES:
Frequency of poor GDS at 1 month after CO exposure between early group and case 1 group in the matched cohort | At 1 month after CO exposure
  Frequency of poor GDS outcome at 1 month after CO exposure between early group and case 1 group
Frequency of poor GDS at 1 month after CO exposure between early group and case 2 group in the matched cohort | At 1 month after CO exposure
  Frequency of poor GDS outcome at 1 month after CO exposure between early group and case 2 group
Frequency of poor GDS at 1 month after CO exposure between case 1 group and case 2 group in the matched cohort | At 1 month after CO exposure
  Frequency of poor GDS outcome at 1 month after CO exposure between case 1 group and case 2 group
Frequency of poor GDS at 6 months after CO exposure between early group and case 1 group in the matched cohort | At 6 months after CO exposure
  Frequency of poor GDS outcome at 6 months after CO exposure between early group and case 1 group
Frequency of poor GDS at 6 months after CO exposure between early group and case 2 group in the matched cohort | At 6 months after CO exposure
  Frequency of poor GDS outcome at 6 months after CO exposure between early group and case 2 group
Frequency of poor GDS at 6 months after CO exposure between case 1 group and case 2 group in the matched cohort | At 6 months after CO exposure
  Frequency of poor GDS outcome at 6 months after CO exposure between case 1 group and case 2 group
The association or trend of change in GDS score at 1 month according to the change of the start time of HBO2 in the overall matched cohort | At 1 month after CO exposure
  The association or trend of change in GDS score at 1 month according to the change of the start time of HBO2 in patients treated with HBO2 within 24 h
The association or trend of change in GDS score at 6 months according to the change of the start time of HBO2 in the overall matched cohort | At 6 months after CO exposure
  The association or trend of change in GDS score at 6 months according to the change of the start time of HBO2 in patients treated with HBO2 within 24 h
Frequency of poor GDS at 1 month after CO exposure in mild CO poisoned patients in the matched cohort | At 1 month after CO exposure
  Frequency of poor GDS outcome at 1 month after CO exposure between early group and late group in mild CO poisoned patients
Frequency of poor GDS at 6 months after CO exposure in mild CO poisoned patients in the matched cohort | At 6 months after CO exposure
  Frequency of poor GDS outcome at 6 months after CO exposure between early group and late group in mild CO poisoned patients
Frequency of poor GDS at 1 month after CO exposure in severe CO poisoned patients in the matched cohort | At 1 month after CO exposure
  Frequency of poor GDS outcome at 1 month after CO exposure between early group and late group in severe CO poisoned patients
Frequency of poor GDS at 6 months after CO exposure in severe CO poisoned patients in the matched cohort | At 6 months after CO exposure
  Frequency of poor GDS outcome at 6 months after CO exposure between early group and late group in severe CO poisoned patients

CONTACTS AND LOCATIONS:
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

REFERENCES:
- [Derived] Lee Y, Cha YS, Kim SH, Kim H. Effect of Hyperbaric Oxygen Therapy Initiation Time in Acute Carbon Monoxide Poisoning. Crit Care Med. 2021 Oct 1;49(10):e910-e919. doi: 10.1097/CCM.0000000000005112. PMID 34074856